CLINICAL TRIAL: NCT03385928
Title: STOP-MSU: Stopping Haemorrhage With Tranexamic Acid for Hyperacute Onset Presentation Including Mobile Stroke Units. A Phase II Randomised, Placebo-controlled, Investigator-driven Trial of Tranexamic Acid Within 2 Hours of Intracerebral Haemorrhage
Brief Title: STOP-MSU: Stopping Haemorrhage With Tranexamic Acid for Hyperacute Onset Presentation Including Mobile Stroke Units
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuroscience Trials Australia (Other)
Collaborators: The Florey Institute of Neuroscience and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTA1702
Record Dates: First submitted 2017-12-13; First posted 2017-12-29 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Intracerebral Haemorrhage
Keywords: ICH; Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Tranexamic Acid; Antifibrinolytic Agents; Fibrin Modulating Agents; Pharmacologic Actions; Cardiovascular Agents; Therapeutic Uses; Hematologic Agents; Hemostatics; Contrast Media; Angiography; Cerebral Angiography; Tomography, X-Ray Computed
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Tranexamic Acid; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study is a prospective phase II randomised, double-blind, placebo-controlled, investigator-driven trial in acute intracerebral haemorrhage patients. The study has 2 arms with 1:1 randomisation to either intravenous tranexamic acid or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Active Comparator): Intravenous tranexamic acid 1000 mg in 100 mL 0.9% NaCl (or in 50ml syringe with 0.9% NaCl) over 10 minutes followed by 1000 mg in 500 mL 0.9% NaCl infusion over 8 hours.
  Interventions: Drug: Tranexamic Acid
- Normal Saline (0.9% NaCl) (Placebo Comparator): 100 mls (or in 50ml syringe) intravenous 0.9%NaCl over 10 minutes followed by 500 ml intravenous 0.9% NaCl infusion over 8 hours.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid — Investigational product given within 2 hours of symptom onset
  Arms: Tranexamic acid
Drug: Normal saline — Placebo given within 2 hours of symptom onset
  Other Names: 0.9%NaCl
  Arms: Normal Saline (0.9% NaCl)

SUMMARY:
The study is a prospective phase II randomised, double-blind, placebo-controlled investigator-driven trial in acute intracerebral haemorrhage patients. The study has 2 arms with 1:1 randomisation to either intravenous tranexamic acid or placebo and will test the hypothesis that in patients with spontaneous ICH, treatment with tranexamic acid within 2 hours of onset will reduce haematoma expansion compared to placebo.

DETAILED DESCRIPTION:
The trial will include patients with acute spontaneous ICH, who are ≥18 years of age and are eligible for treatment within 2 hours of stroke onset. A sample size of 326 patients is calculated to give 80% power to detect a large effect size assuming mean relative ICH haematoma growth of 38% in the placebo arm compared to 19% in the active treatment arm and standard deviation of 19%, inflated for nonparametric analysis. Adaptive increase in sample size will be performed if the result of interim analysis of the first 144 patients is promising, using the methodology of Mehta and Pocock. The maximum sample size is capped at 326. Standard CT for initial diagnosis of suspected stroke patients will be performed. Neurological impairment and functional scores will be measured by a neurologist or health care professional trained in their administration. The assessors will be blinded to the treatment group. Patients eligible for the RCT will be randomised in a 1:1 ratio to receive either tranexamic acid or placebo stratified by treating centre and utilising randomly permuted blocks of random size.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with an acute ICH
2. Age ≥18 years
3. Treatment can commence within 2 hours of symptom onset (or in patients with unknown time of symptom onset, the time patient was last known to be well)
4. Consent can be obtained from participant or person responsible. When emergency treatment procedures have been followed the participant or person responsible will be asked for consent to continue in the study.

Exclusion Criteria:

1. Glasgow coma scale (GCS) total score of <8
2. Brainstem ICH
3. ICH volume >70 ml as measured by the ABC/2 method
4. ICH known or suspected by study investigator to be secondary to trauma, aneurysm, vascular malformation, haemorrhagic transformation of ischaemic stroke, cerebral venous thrombosis, thrombolytic therapy, tumour, or infection
5. Any history or current evidence suggestive of venous or arterial thrombotic events within the previous 12 months, including clinical, ECG, laboratory, or imaging findings. Clinically silent chance findings of old ischemia are not considered exclusion.
6. Hereditary or acquired haemorrhagic diathesis or coagulation factor deficiency.
7. Use of heparin, low-molecular weight heparin, GPIIb/IIIa antagonist, or oral anticoagulation (e.g. warfarin, factor Xa inhibitor, thrombin inhibitor) within the previous 72 hours.
8. Pregnancy (women of childbearing potential must be tested)
9. Planned surgery for ICH within 24 hours
10. Concurrent or planned treatment with haemostatic agents (e.g. prothrombin complex concentrate, vitamin K, fresh frozen plasma, or platelet transfusion)
11. Participation in any investigational study in the last 30 days
12. Known terminal illness or planned withdrawal of care or comfort care measures
13. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Haematoma growth by 24±6 hours as defined by either ≥33%or ≥6ml increase from baseline ICH volume (mls) | 24 hours(plus or minus 6 hours)
  Relative ICH haematoma growth

SECONDARY OUTCOMES:
Haematoma growth by 24±6 hours as defined by ≥33%or ≥6ml increase from baseline in intracerebral haematoma volume, or any increase intraventricular haematoma volume | 24 hours ±6 hours
  ICH or IVH growth at 24 hours ±6 hours from baseline
Absolute haematoma growth by 24±6 hours | 24 hours ±6 hours
  ICH growth as defined by either ≥33%or ≥6ml increase from baseline from baseline, adjusted for baseline ICH volume
Relative haematoma growth by 24±6 hours | 24 hour ±6 hours
  Relative ICH growth volume, adjusted for baseline ICH volume
Absolute intraventricular haematoma growth by 24 hours ±6 hours | 24 hours ±6 hours
  IVH growth at 24 hours ±6 hours from baseline
Absolute intracerebral plus intraventricular haematoma growth by 24±6 hours | 24 hours ±6 hours
  ICH plus IVH growth from baseline
The number of patients with mRS 0-3 or back to pre-stroke level at 3 months | 90 days ± 7 days
  mRS 0-3 or back to pre-stroke level at 3 months
The number of patients with mRS 0-4 or back to pre-stroke level at 3 months | 90 days ± 7 days
  mRS 0-4 or back to pre-stroke level at 3 months
Categorical shift in mRS at 3 months | 90 days ± 7 days
  mRS 0-4 or back to pre-stroke level, or mRS 0-3 or back to pre-stroke level (with lowest mRS score being the better outcome)
Major thromboembolic events (myocardial infarction, ischaemic stroke, or pulmonary embolism) within 3 months | 3 months from baseline
  Safety outcome
Death within 3 months | 3 months from baseline
  Safety outcome
Death within 7 days | 7 days from baseline
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Donnan, MD, Principal Investigator — The Florey Institute of Neuroscience and Mental Health; Stephen Davis, MD, Principal Investigator — Melbourne Health Dept of Neurology & The University of Melbourne Dept of Medicine; Henry Zhao, MD, Principal Investigator — Melbourne Health Dept of Neurology & The University of Melbourne Dept of Medicine
Locations (25):
- Australia (15):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Mobile Stroke Unit, Parkville, Victoria
- Helsinki University Hospital, Helsinki, Finland
- New Zealand (3):
  - CDHB Christchurch Hospital, Christchurch
  - Palmerston North Hospital, Palmerston North
  - Wellington Hospital, Wellington
- Taiwan (3):
  - E-DA Hospital, Kaohsiung City, Yanchao District
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Vietnam (3):
  - Bach Mai Hospital, Hanoi
  - Military 103 Hospital, Hanoi
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City

REFERENCES:
- [Derived] Yassi N, Zhao H, Churilov L, Wu TY, Ma H, Nguyen HT, Cheung A, Meretoja A, Mai DT, Kleinig T, Jeng JS, Choi PMC, Duc PD, Brown H, Ranta A, Spratt N, Cloud GC, Wang HK, Grimley R, Mahawish K, Cho DY, Shah D, Nguyen TMP, Sharma G, Yogendrakumar V, Yan B, Harrison EL, Devlin M, Cordato D, Martinez-Majander N, Strbian D, Thijs V, Sanders LM, Anderson D, Parsons MW, Campbell BCV, Donnan GA, Davis SM; STOP-MSU Trial Investigators. Tranexamic acid versus placebo in individuals with intracerebral haemorrhage treated within 2 h of symptom onset (STOP-MSU): an international, double-blind, randomised, phase 2 trial. Lancet Neurol. 2024 Jun;23(6):577-587. doi: 10.1016/S1474-4422(24)00128-5. Epub 2024 Apr 20. PMID 38648814
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112